CLINICAL TRIAL: NCT02918045
Title: Dental Extractions in Patients Under Dual Antiplatelet Therapy: Comparison of Two Local Hemostatic Techniques
Brief Title: Dental Extractions in Patients Under Dual Antiplatelet Therapy
Acronym: DUALex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Bruno Guardieiro, PhD degree student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DUALex
Record Dates: First submitted 2016-09-21; First posted 2016-09-28 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Blood Coagulation Disorders
Keywords: Tooth Extraction; Surgical Hemostasis; Platelet Aggregation Inhibitors; Chitosan
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind, Randomized, Split-mouth
Who Masked: Participant
Masking Description: The participant (patient) does not know which site received the study local hemostatic or the control local hemostatic.It is not possible for the surgeon to be blinded in this case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hemcon Dental Dressing (Experimental): The HemCon® Bandage is an FDA-cleared chitosan-based flat bandage that controls severe arterial bleeding from traumatic injuries. In comparison to traditional bandages, the HemCon® Bandage provides superior control of bleeding, wound site adhesiveness, multiple injury site usage, biocompatibility and provides a barrier to infective agents.
  Interventions: Device: HemCon Dental Dressing
- Oxidized Cellulose Gauze (Active Comparator): A common hemostatic measure after dental extractions involves the placement of an absorbable oxidized cellulose gauze Surgicel (Ethicon, Inc, San Angelo, TX) into the extraction socket. This treatment was chosen as the study control to compare the HemCon Dental Dressing to the standard local hemostatic care for oral surgery subjects.
  Interventions: Device: Oxidized Cellulose Gauze

INTERVENTIONS:
Device: HemCon Dental Dressing — The Hemcon Dental Dressing is an oral wound dressing made of chitosan.
  Arms: Hemcon Dental Dressing
Device: Oxidized Cellulose Gauze — A common hemostatic measure after dental extractions placed into the extraction socket.
  Other Names: Surgicel (Ethicon, Inc, San Angelo, TX)
  Arms: Oxidized Cellulose Gauze

SUMMARY:
The purpose of this study is to compare two hemostatic agents in patients under dual antiplatelet therapy using the intraoral bleeding time after dental extractions.

DETAILED DESCRIPTION:
Postoperative hemostasis is a fundamental patient management issue in the oral and maxillofacial surgery setting. The risk of excessive bleeding prompts physicians to stop multiple antiplatelet agents before minor surgery, which puts coronary stenting patients at risk for adverse thrombotic events. Adequate hemostasis must be achieved in order to make oral surgeries possible for these patients without discontinuation of the antiplatelet regimen. The HemCon Dental Dressing (HemCon Medical Technologies, Inc, Beaverton, OR) is a novel chitosan-based hemostatic agent which may greatly improve upon the efficacy of wound healing and hemostasis both in extent and time for minor oral surgeries. Dental extractions will be performed in patients under dual antiplatelet therapy without altering their medication regimen. All patients will require to have two or more surgical sites so they will have internal surgical control sites. Cutaneous bleeding time and platelet aggregation tests will be obtained prior to extractions. The primary hemostasis will be evaluated by measuring the intraoral bleeding time after each extraction and further bleeding and healing outcomes will be ascertain by phone questionaires and clinical evaluations. The aim of this study is to evaluate the effectiveness of HemCon Dental Dressing in controlling post extraction bleeding and to ascertain its role in healing of extraction wounds compared to a standard haemostasis method.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring two or more dental extraction procedures.
* Patients must be under dual antiplatelet therapy of any kind.
* Patients must be 18 years of age or older.
* Patients must be available for a minimum of one post operative evaluation to be scheduled at the time of the procedure approximately 7 days post surgery.
* Extraction sites do not require primary closure of suturing.
* Willingness and ability to provide informed consent

Exclusion Criteria:

* Patients who are currently undertaking other anticoagulant medications (e.g., aspirin, coumadin, heparin) or have discontinued their anticoagulant medications.
* History of heart attack in less than 1 week.
* Patients with seafood allergy.
* Unable of unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Primary bleeding | Intraoperative
  Primary bleeding will be evaluated by recording the intra-oral bleeding time. The extraction site will be observed for 2 min without gauze in place. At the end of 2 min, gauze is placed over the extraction site to remove blood extending beyond the tooth socket. After blotting the extraction site, any bleeding that extends beyond the crest of the socket will be recorded as a positive test result (i.e., onto surrounding gingival tissues) during an observation period of 1 min. This same procedure was performed at 5, 8, 11, 14, and 20 min after the extraction. Intra-oral bleeding time is defined as the length of time for bleeding to cease to extend beyond the tooth socket.

SECONDARY OUTCOMES:
Point-of-care platelet function test | Day before dental extraction
  Blood platelet function plays a pivotal role in hemostasis during surgery and following traumatic injuries. The ability to assess platelet function before the intervention is desirable in patients undergoing dental extraction procedures. A point-of-care platelet function test (Multiplate - Roche Diagnostics, Mannheim, Germany) will be performed the morning before dental extraction to assess platelet function inhibition due to dual antiplatelet therapy.

OTHER OUTCOMES:
Secondary bleeding (T1) | 10-15 hours after dental extraction
  Secondary bleeding (T1) will be evaluated by telephone with standardized questionnaire including the following: whether bleeding occurred after the individual left the dental clinic (y/n); whether gauze was needed to be placed due to bleeding (y/n); and whether an emergency service or dental clinic was visited due to bleeding (y/n).
Secondary bleeding (T2) | 45-50 hours after dental extraction
  Secondary bleeding (T2) will be evaluated by telephone with standardized questionnaire including the following: whether bleeding occurred after the individual left the dental clinic (y/n); whether gauze was needed to be placed due to bleeding (y/n); and whether an emergency service or dental clinic was visited due to bleeding (y/n).
Intra patient healing comparison | 1 week post surgery
  Healing will be compared between the study and control sites and assessed on a scale of 1-3 with 1 representing the healing of the study site being significantly worse than the control; 2 representing the healing of the study site being the same as the control, and 3 meaning the healing of the study site was significantly better than the control.

CONTACTS AND LOCATIONS:
Overall Officials: Itamara LI Neves, PhD, Principal Investigator — University of Sao Paulo; José C Nicolau, PhD, Study Director — University of Sao Paulo
Locations (1):
- Instituto do Coração (InCor HCFMUSP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided